CLINICAL TRIAL: NCT04784923
Title: Detecting Malposition of Trans-pedicle Screw From AP and LAT Plain Radiographs
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: N202007008
Record Dates: First submitted 2021-02-22; First posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2020-06

CONDITIONS: Orthopedics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Instrumentation patients: Instrumentation patients

SUMMARY:
Our study focuses on reducing the use of CT (Computer Tomography) for pedicle screw instrumentation, replacing CT with X-ray. We are writing a program to measure the position on X-ray seeing whether the position meets that on CT after operation. In the future,our method can be used in fluoroscopy, helping us detecting screw malposition efficiently during the surgeries, and hoping reduce complications.

DETAILED DESCRIPTION:
Most of the spine surgeries are decompression, fusion, with instrumentation.Instrumentation needs screws. Pedicle screws are often used. If the pedicle screws are mal-located, that is breaking the pedicle wall; the consequence may be injury of the spinal cord, or nerve root. Some lucky patients may have no symptom; however, broken pedicle will reduce the fixation strength which may reduce fusion rate.

Detecting malposition screws, currently we use CT (computer tomography) method. The surgeon carefully read the CT slice by slice, looking for clues of screws malposition. However, CT is costly both price and radiation dose.We invented a plain radiograph method which has been pilot tested in one patient with good correction rate. The purpose of this study is to solve the following two clinical problems:

1. What are the inter-observer and intra-observer reliabilities of CT method?
2. The radiation dose for CT method is too high. Does our plain radiograph method has the same correction rate? Materials and methods We planned to collect about 100 patients received spinal fusion and instrumentation who has preoperative CT(or MRI) and postoperative plain radiographs and CT. We will firstly verify CT method's reproducibility by interobserver and intra-observer reliability test. With the same databank, we will use our plain radiograph method again, and test if the two methods' results are the same by Chi-square test.

Conclusion:

We hope our study can reduce some unnecessary CT examination. In the future,our method can be used in fluoroscopy, helping us detecting screw malposition efficiently during the surgeries, and hoping reduce complications.

ELIGIBILITY:
Inclusion Criteria:

* s/p pedicle screw insertion surgery
* good quality postoperative plain radiograph
* good quality postoperative CT

Exclusion Criteria:

* poor quality postoperative plain radiograph
* poor quality postoperative CT

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from Shuang Ho Hospital
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Verify the position of pedicle screw on X-ray compared to that on CT's | 30 days
  Investigators will verify CT method's reproducibility by interobserver and intra-observer reliability test. With the same databank, investigators will use the plain radiograph method again, and test if the two methods' results are the same by Chi-square test.

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Kun Liaw, Study Chair — Taipei Medical University

IPD SHARING:
Plan to Share IPD: Undecided